CLINICAL TRIAL: NCT06435637
Title: Collagen Digestion and Amino Acid Absorption Kinetics and the Effect on Muscle & Skin
Brief Title: Effects of Ingesting Multiple Boluses of Collagen on Muscle & Skin Connective Protein Synthesis in Vivo in Humans
Acronym: CODIAK
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: METC 22-018
Record Dates: First submitted 2024-04-22; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Muscle Protein Synthesis
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Double-blind, parallel-group, placebo-controlled intervention study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen protein (Experimental): 100 g of collagen peptides (in boluses) with vitamin C
  Interventions: Dietary Supplement: Collagen protein; Behavioral: Resistance exercise
- Placebo (Placebo Comparator): Non-caloric placebo (flavoured water) drinks, with vitamin C.
  Interventions: Behavioral: Resistance exercise

INTERVENTIONS:
Dietary Supplement: Collagen protein — Ingestion of 40, 20, 20 and 20 gram of collagen protein right after and every 2 hours after a bout of exercise
  Arms: Collagen protein
Behavioral: Resistance exercise — A single resistance exercise session of the leg press and leg extension exercise

SUMMARY:
Rationale: Collagen protein is the central structural component of extracellular connective tissues within skeletal muscle, bone, cartilage and skin. Dietary collagen peptides are a promising protein source to deliver the specific amino acid precursors required to support an increase in connective tissue protein synthesis across several tissues (e.g. muscle, skin). However, the digestion and absorption kinetics of multiple boluses of collagen peptides and the subsequent impact on muscle and skin connective tissue protein synthesis rates have not yet been assessed in vivo in humans.

Objective: To assess the impact of ingestion of multiple boluses of collagen peptides on muscle connective and skin protein synthesis in vivo in humans.

Study design: Double-blind, parallel-group, placebo-controlled intervention study.

Study population: 20 healthy young males, aged 18-35 years.

Intervention : Participants will perform unilateral resistance exercise followed by the ingestion of either 100 g of collagen peptides (in boluses) or a non-caloric placebo (flavoured water) drinks, while all drinks will contain vitamin C. Continuous intravenous stable isotope amino acid tracer infusions will be applied, plasma, skin and muscle samples will be collected in order to assess protein synthesis rates in skin and muscle tissue.

Main study parameters/endpoints: Primary study parameters are muscle connective protein synthesis rates. Secondary study parameters are skin and myofibrillar protein synthesis rates, plasma amino acid concentrations and body composition.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-35 years
* Male
* Healthy, recreationally active (participating in recreational sports activities ≥ 1 and ≤ 6 h per week, with a maximum of 2 h resistance-type exercise)
* 18.5 ≤ BMI ≤ 30 kg/m2
* No physical limitations (i.e. able to perform all activities associated with daily living in an independent manner).

Exclusion Criteria:

* Female
* Smoking
* Musculoskeletal disorders
* Metabolic disorders
* Use of any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescribed acne medications).
* Chronic use of gastric acid suppressing medication or anti-coagulants
* Unstable weight over the last three months
* Diagnosed GI tract disorders or diseases
* Blood donation in the past 2 months

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Muscle connective protein synthesis rates rested leg | one value calculated over 8 hours
  The primary analysis will be an independent t-test, comparing postprandial muscle connective protein synthesis rates over the 0-8 h period (i.e., one integrated value) in the rested condition between groups.

SECONDARY OUTCOMES:
Muscle connective protein synthesis rates exercised leg | one value calculated over 8 hours
  Independent t-test, comparing postprandial muscle connective protein synthesis rates over the 0-8 h period (i.e., one integrated value) in the exercised condition between groups.
Myofibrillar protein synthesis rates rested leg | one value calculated over 8 hours
  Independent t-test, comparing postprandial myofibrillar protein synthesis rates over the 0-8 h period (i.e., one integrated value) in the rested condition between groups.
Myofibrillar protein synthesis rates exercised leg | one value calculated over 8 hours
  Independent t-test, comparing postprandial myofibrillar protein synthesis rates over the 0-8 h period (i.e., one integrated value) in the exercised condition between groups.
Skin protein synthesis rates | one value calculated over 8 hours
  Independent t-test, comparing postprandial skin protein synthesis rates over the 0-8 h period (i.e., one integrated value).
Plasma insulin concentrations | measured over the 8 hour post-prandial period
  Plasma insulin concentrations
Plasma amino acids concentrations | measured over the 8 hour post-prandial period
  Plasma amino acids concentrations

OTHER OUTCOMES:
Age | baseline
  age in years
Dietary macronutrient intake | 2 days before test days
  assessed by written dietary intake records
Body mass | baseline
  body mass in kg
Height | baseline
  Height in m
Lean mass | baseline
  Measured by DXA
One repetition maximum of the legs | baseline
  maximum strength of both legs

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided